CLINICAL TRIAL: NCT00721643
Title: Absorption Kinetics of Polyphenols in Angel's Plant (Angelica Keiskei)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Kyung-Jin Yeum, Scientist, Jean Mayer USDA-Human Nutrition Research Center on Aging at Tufts University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HNRCA2580; BioGreen 20070301034009
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Oxidative Stress
Keywords: Angelica keiskei; absorption kinetics; quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Healthy control, 5g dry power of angel's plant (Angelica keiskei)
  Interventions: Dietary Supplement: angel's plant (Angelica keiskei)
- 2 (Experimental): Metabolic syndrome, 5g dry powder of angel's plant (Angelica keiskei)
  Interventions: Dietary Supplement: Angel's plant (Angelica keiskei)

INTERVENTIONS:
Dietary Supplement: angel's plant (Angelica keiskei) — Healthy control, one time dose of 5g dry power of Angelica keiskei
  Arms: 1
Dietary Supplement: Angel's plant (Angelica keiskei) — Metaboic syndrome subjects, one time dose of 5g dry powder of angel's plant (Angelica keiskei)
  Arms: 2

SUMMARY:
The absorption kinetics of polyphenols in angel's plant (Angelica keiskei), which is a dark green leafy vegetable rich in antioxidant nutrients, will be determined in older adults in this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (>60 yr, n=5)
* subjects with metabolic syndrome (>60 yr, n=5)
* Subjects who has

  * high fasting plasma glucose (>5.6 mmol/L),
  * central obesity (waist-hip ratio, >0.9 for men, >0.85 for women)
  * either high blood pressure (>130/85 mmHg) or high triacylglycerol (>1.7 mmol/L) will be selected to have metabolic syndrome.
* normal hematological parameters, normal serum albumin, normal liver function, and normal kidney function
* no history of smoking or alcoholism.

Exclusion Criteria:

* consume >7 alcoholic drinks/wk
* taking cholesterol medication or hormone replacement

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Plasma quercetin | 0, 30, 60, 100, 180, 240, 300, 360, 420 & 480 min

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Jin Yeum, Ph.D., Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA-Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States